CLINICAL TRIAL: NCT04255576
Title: A Phase Ib/II, Multicenter, Single-Arm, Open-Label Study to Evaluate the Efficacy and Safety of JMT103 in Surgically Unsalvageable or Refractory Giant Cell Tumor of Bone
Brief Title: Efficacy and Safety of JMT103 in Patients With Giant Cell Tumor of Bone
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMT103CN03
Record Dates: First submitted 2020-01-13; First posted 2020-02-05 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Giant Cell Tumor of Bone
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: JMT103 (Experimental): Eligible subjects will receive JMT103 at a dose of 2 mg/kg SC Q4W with a loading dose of 2 mg/kg SC on study days 8 and 15.
  Interventions: Dietary Supplement: Dietary Supplement: Calcium/Vitamin D

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Calcium/Vitamin D — All subjects should be adequately supplemented with calcium and vitamin D (at least 500 mg of calcium and 400 IU of vitamin D), except in the case of pre-existing hypercalcemia.

SUMMARY:
This is a phase Ib/II, multicenter, single-arm, open-label study to evaluate the efficacy and safety of JMT103 in patients with surgically unsalvageable or refractory giant cell tumor of bone (GCTB).

DETAILED DESCRIPTION:
The objective of the trial is to evaluate the efficacy and safety of JMT103 in patients with GCTB that is surgically unsalvageable or for which the planned surgery is associated with severe morbidity.

This study consists of two parts (phase Ib and II). In the phase Ib part, 6 to 12 subjects will be enrolled, and the safety, pharmacokinetics and pharmacodynamics of JMT103 will be evaluated after treatment for more than 4 weeks. And then the phase II part will be conducted, in which, 125 subjects will be enrolled.

Eligible subjects will receive JMT103 at a dose of 2mg/kg subcutaneously (SC) every 4 weeks (Q4W) with a loading dose of 2mg/kg SC on study days 8 and 15 until disease progression, tumor resection (the pathologic outcome after surgical resection is CR or PR), intolerable toxicity, decision by the participant to discontinue, or decision by the investigator that the subject could no longer benefit from the treatment (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed and signed informed consent.
2. Male or female, Adults, 18 years and older
3. Histologically confirmed GCTB that is surgically unsalvageable or for which the planned surgery is associated with severe morbidity.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

Exclusion Criteria:

1. Fertile subjects refuse to use effective contraception methods from the signing of the informed consent to 6 months after the last dose;
2. Active dental or jaw condition which requires oral surgery, including tooth extraction;
3. Currently receiving other anti-tumor therapy (radiotherapy, chemotherapy or arterial embolization, etc.);
4. Concurrent treatment with bisphosphonates;
5. Known history of second malignancy within the past 5 years, except for basal cell carcinoma or cervical carcinoma in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Giant Cell Tumor Response | From enrollment until 12 weeks
  A treatment response was defined for participants with tissue samples obtained and measured by histopathology as: at least 90% elimination of giant cells relative to Baseline. A response was defined for participants who have only radiographs (histopathology not available) as lack of progression of the target lesion (PR or CR) at week 12 by radiographic measurements compared with Baseline.

SECONDARY OUTCOMES:
Proportion of Participants with Adverse Events (AEs) | From enrollment until 90 days after the last dose
Objective Response Rate (ORR) | From enrollment until the last dose, no more than 24 months
Changes in Brief Pain Inventory Short Form (BPI-SF) | From enrollment until the last dose, no more than 24 months
  Assess pain and its effects on patients' mood, sleep, ability to move, appetite, daily life, ability to walk, and social interaction
Percentage of Patients with Surgical Resection of Tumor | From enrollment until the last dose, no more than 24 months
Serum JMT103 Trough Concentrations | From enrollment until 90 days after the last dose
Percent Change from Baseline in Serum C-terminus Peptide (of Type 1 Collagen) and Urinary N-telopeptide Corrected for Urine Creatinine | From enrollment until the last dose, no more than 24 months
Number of Participants with Anti-JMT103 Antibodies | From enrollment until 90 days after the last dose
Disease Control Rate (DCR) | From enrollment until the last dose, no more than 24 months
Time to Progress (TTP) | From enrollment until the last dose, no more than 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ji Shui Tan Hospital, Beijing, China

REFERENCES:
- [Derived] Xu H, Zhou Y, Wei F, Ding Y, Shan H, Yang Y, Liu W, Jin T, Luo Y, Tang F, Lu M, He X, Zhang W, Yang S, Zhang L, Wang J, Li H, Tu C, Niu X. JMT103 versus Non-Denosumab or Denosumab Treatment in Chinese Patients with Unresectable or Surgically Challenging Giant Cell Tumor of Bone: A Propensity Score-Matched Comparison. Cancer Med. 2025 Nov;14(22):e71340. doi: 10.1002/cam4.71340. PMID 41292259
- [Derived] Xu H, Zhou Y, Liang L, Shen J, Yan W, Wang J, Li J, Zhang X, Huang G, Bi W, Guo Z, Xiao Y, Lin J, Yao W, Tong Z, Zhou W, Zhang G, Ye Z, Wang D, Yang J, Fan Z, Liu C, Qu G, Zhang Q, Wei F, Liu W, Tu C, Li H, Yuan J, Niu X. Efficacy and safety of JMT103 in patients with unresectable or surgically-challenging giant cell tumor of bone: a multicenter, phase Ib/II study. Nat Commun. 2024 Nov 5;15(1):9541. doi: 10.1038/s41467-024-53686-4. PMID 39500883